CLINICAL TRIAL: NCT05926076
Title: Comparative Study of COVID-19 Infection in Renal Transplant Recipients and Non Transplant Recipients
Brief Title: COVID-19 Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin First Central Hospital (Other)
Collaborators: Shenzhen Third People's Hospital (Other)
Responsible Party: Principal Investigator, Yingxin FU.MD, Head of department, Tianjin First Central Hospital
Other Study IDs: 2023-036-02
Record Dates: First submitted 2023-06-24; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: COVID-19; Renal Transplant Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kidney Transplant Recipients Group (KTR)
  Interventions: Other: Treatment plan
- Non-Kidney Transplant Recipients Group（NKTR）
  Interventions: Other: Treatment plan

INTERVENTIONS:
Other: Treatment plan — Patients with different diagnoses will get different treatment options

SUMMARY:
Post-transplant patients with COVID-19 infection who attended Shenzhen No. 3 Hospital from December 2022 to February 2023, and enrolled the general population with COVID-19 infection who were hospitalized during the same period, matched by age and gender.

DETAILED DESCRIPTION:
Data collection：Age, BMI, underlying comorbidities and other basic information were collected retrospectively from the two groups. The medical records were used to collect information about the patients' new coronavirus infection, such as the time of onset of symptoms, time of diagnosis, time of conversion and common symptoms such as fever, cough, nasal congestion and runny nose, muscle aches and pains.To compare the differences of the diagnosis and treatment of KTRs and the general population infected with Omicron

ELIGIBILITY:
Inclusion Criteria:

Confirmed novel coronavirus infection between December 2022 to February 2023,

Exclusion Criteria:

Age less than 18; failure of the transplanted kidney before the new coronavirus infection; exclusion of oral immunosuppressed and other types of organ transplant recipients from the non-renal transplant population

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: post-transplant patients with COVID-19 infection who attended Shenzhen No. 3 Hospital from December 2022 to February 2023, and enrolled the general population with COVID-19 infection who were hospitalized during the same period, matched by age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 610 (Estimated)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
ICU admission or death | through study completion, an average of 1 month
  patients have ICU admission or death

CONTACTS AND LOCATIONS:
Locations (1):
- yingxin Fu, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No